CLINICAL TRIAL: NCT06664398
Title: Preventive Effects of Different Volumes of High-Intensity Interval Training on Risk Factors for Metabolic Syndrome in Overweight Young Women
Brief Title: Preventive Effects of Different Volumes of High-Intensity Interval Training on Risk Factors for MS in Overweight Young Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sport University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PEDVHIITRFMOYW
Record Dates: First submitted 2024-10-28; First posted 2024-10-29 (Actual); Last update posted 2024-10-29 (Actual); Status verified 2024-10

CONDITIONS: Metabolic Syndrome
Keywords: high-intensity interval training; overweight; metabolic syndrome; risk factor; prevention
MeSH Terms: conditions — Metabolic Syndrome; Overweight

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- 1HIIT group (Active Comparator)
  Interventions: Behavioral: one HIIT
- 4HIIT group (Active Comparator)
  Interventions: Behavioral: four HIIT
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: one HIIT — one HIIT high intensity interval training
  Arms: 1HIIT group
Behavioral: four HIIT — four HIIT high intensity interval training
  Arms: 4HIIT group

SUMMARY:
This study investigates the effects of different volumes of high-intensity interval training on risk factors for metabolic syndrome in overweight young women.

DETAILED DESCRIPTION:
The sedentary and inactive female overweight subjects, aged 18 to 30 years, were randomly divided into three groups: high volume high-intensity interval training group (4HIIT group), low volume high-intensity interval training group (1HIIT group) and control group (CON group). Human morphological measures, blood pressure, insulin resistance, blood analysis, and cardiorespiratory fitness were measured at baseline and after exercise intervention.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-30 years;
* BMI≥24kg/m2, indicating overweight and high risk of metabolic syndrome;
* Maintaining a stable body weight for the three months prior to the study.

Exclusion Criteria:

* Regular participation in physical exercise (≥3 times/week, exercise time≥30min/time);
* Any respiratory, musculoskeletal, or cardiovascular diseases;
* Medical or other contraindications for exercise;
* Taking medications that affect metabolism;
* Smoking and/or drinking habits.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Weight | 8 weeks
  Changes in Weight before and after intervention.
Body Mass Index (BMI) | 8 weeks
  Changes in BMI before and after intervention.
body fat percentage | 8 weeks
  Changes in body fat percentage before and after intervention.
waist circumference (WC) | 8 weeks
  Changes in WC before and after intervention.
Systolic blood pressure (SBP) | 8 weeks
  Changes in SBP before and after intervention.
Diastolic blood pressure (DBP) | 8 weeks
  Changes in DBP before and after intervention.
Fasting plasma glucose (FPG) | 8 weeks
  Changes in FPG before and after intervention.
Triglyceride (TG) | 8 weeks
  Changes in TG before and after intervention.
High-density lipoprotein cholesterol (HDL-C) | 8 weeks
  Changes in HDL-C before and after intervention.

SECONDARY OUTCOMES:
Non high-density lipoprotein cholesterol (Non HDL-C) | 8 weeks
  Changes in HDL-C before and after intervention.
Insulin | 8 weeks
  Changes in insulin before and after intervention.
Homeostatic model assessment for insulin resistance (HOMA-IR) | 8 weeks
  12、Homeostatic model assessment for insulin resistance (HOMA-IR) Changes in HOMA-IR before and after intervention.
Triglyceride-glucose (TyG) index | 8 weeks
  Changes in TyG index before and after intervention.
Triglyceride-to-high density lipoprotein cholesterol ratio (TG/HDL-C ratio) | 8 weeks
  Changes in TG/HDL-C ratio before and after intervention.
Visceral fat area (VFA) | 8 weeks
  Changes in VFA before and after intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Sports Medicine and Rehabilitation, Beijing Sport University, Beijing, China